CLINICAL TRIAL: NCT04105712
Title: The Biobehavioral Impact of Diet Quality on Affect and Craving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Ashley Gearhardt, Associate Professor of Psychology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00156725
Record Dates: First submitted 2019-09-23; First posted 2019-09-26 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Food Addiction; Withdrawal
Keywords: withdrawal; highly processed food; food addiction
MeSH Terms: conditions — Food Addiction

STUDY DESIGN:
Intervention Model Description: Multi-method, within subjects, prospective, experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre and Post Dietary Change (within subjects) (Experimental): Participants do an initial call for baseline data. Then the active assessment period (pre / post dietary change) begins. Pre - dietary change procedure is 5 days of standard high HP diet while completing daily electronic assessments of withdrawal, ecological momentary assessments, and a phone appointment. Post - dietary change is 5 days of lower HP diet (food provided for 3 of 5 days) while completing daily electronic assessments of withdrawal, ecological momentary assessments, and a phone appointment. Daily assessments of affect, craving, and withdrawal are all virtual. On day 4-5 of post assessment, participants complete a food journal to report foods they ate to ensure compliance to low HP food diet. The pre / post-dietary change phone appointments include 1) psychosocial stress task, 2) cue reactivity task, 3) questionnaires 4) self-reported weight. Participants may also complete a follow up period of questionnaires every other day and self-report weight at the end of follow up.
  Interventions: Behavioral: Dietary Change (low in highly processed foods)

INTERVENTIONS:
Behavioral: Dietary Change (low in highly processed foods) — For post-dietary change, food is provided for 3 days (participants provide own food and do food journals the other 2 days to confirm adherence). University of Michigan's Nutrition Obesity Research Center (NORC)'s Metabolic Kitchen prepares the food. Low HP food diet is based on prior methods where participants are placed on an isocaloric diet composed of 5% or less of calories from added sugar and 10% or less of overall calories from total sugar. No foods that meet the criteria for a HP food (defined by Kant and colleagues) that corresponds to: sweeteners (sugar, candy, etc); carbonated and non-carbonated beverages (fruit drinks, sweetened / diet beverages, etc.); baked / dairy desserts (cookies, ice cream, etc.); salted snacks (potato chips, etc.) and fast foods (pizza, cheeseburgers, etc.) are included in diet portions. The overall macro nutrient composition of the diet will be approximately 20-25% of kcal from protein, 30-35% of kcal from fat, and 40-50% of kcal from carbohydrates.

SUMMARY:
The current study experimentally investigates whether reducing highly processed (HP) foods (defined in this study as foods high in added sugars) leads to, psychological and / or behavioral indicators of withdrawal. The following hypotheses are tested:

1. To test the hypothesis that reducing highly processed food intake will result in higher daily reports of physical (e.g. headaches), cognitive (e.g. difficulty concentrating), and affective (e.g., irritability) withdrawal symptoms).
2. To test the hypothesis that reducing highly processed food intake will result in increased negative affect (e.g., irritability, depression) as indicated by and psychological (self - reported distress ratings; daily emotion / mood reports) measures.
3. To test the hypothesis that reducing highly processed food intake will result in increased food craving as indicated by psychological (self - report craving ratings; daily craving report) measures.

All activities are completed remotely. Participants complete 4 phone appointments with a trained member of the research team. Daily questionnaires and ecological momentary assessments are completed at home between phone appointments. The initial call signs electronic consent and gets baseline measurements (questionnaires). After the initial call, participants start an active assessment period (pre / post dietary change assessments). Pre-dietary change includes at home questionnaires and ecological momentary assessments while eating a typical diet. It also includes the second phone appointment. Post-dietary change includes at home questionnaires and ecological momentary assessments while consuming 3 days of food portions lower in highly processed foods. Participants will complete a food journal on the remaining 2 days of post - dietary change assessment to report what food they ate. Post - dietary change also includes the third phone appointment. The second and third phone appointments each include computer tasks and questionnaires. The final phone appointment is a debriefing interview. Participants planning to continue eating a healthier diet may also be invited to complete a follow-up period, which involves answering a short questionnaire at home every other day for two weeks. 7 individuals had in-person data collected prior to the pandemic requiring a shift to virtual data collection.

ELIGIBILITY:
Inclusion Criteria:

* Age 25 to 40
* Access to internet, private computer and smart phone
* Overweight (self-report BMI above 25.0)
* Moderately or Highly motivated to eat a healthier diet
* Mild, moderate or severe levels of addictive like eating (2 or higher on the Yale Food Addiction Scale)
* Fluent in english
* Willing to follow dietary guidelines provided by study team and eat only provide food for 3 days. Willing to delay dietary change until instructed to do so

Exclusion Criteria:

* Use of nicotine in the past month, cannabis in the past month, or illicit drugs in the past 6 months
* Weight fluctuation of 20+ pounds in the last 3 months
* Attempted weight loss using a formal weight loss program (e.g. weight watchers) in the last month
* Prior weight loss surgery (e.g. bariatric surgery)
* Medications or medical conditions that may impact study results such as medications that impact appetite, heart rate, or reward functioning (e.g. taking synthroid or has diabetes)
* Current major psychiatric diagnoses (e.g., bipolar, schizophrenia, substance use disorder, eating disorder)
* A diagnosis of a restrictive eating disorder in the past 5 years (anorexia nervosa, bulimia nervosa, purging disorder)
* Significant dietary restrictions (e.g. allergies, veganism)
* currently pregnant, breastfeeding, trying to get pregnant, or within 6 months of giving birth

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Increase in affective withdrawal symptoms during post-dietary change assessment using the Highly Processed Food Withdrawal Scale (PRoWS). | Through study completion, an average of 1 month
  The PRoWS is a validated self-report measure of indicators of withdrawal. Affective withdrawal symptoms are measured by asking participants to complete the Highly Processed Food Withdrawal Scale (PRoWS), which is a validated self-report measure of withdrawal. PRoWS questions ask about current feelings / emotions. Response options are "strongly disagree" "disagree" "feel neutral" "agree" and "strongly agree". Participants are asked to complete these measures every day of the pre and post dietary change. Change in self - report responses on the PRoWS at pre dietary change compared to post dietary change will be used for analyses.
Increase in negative affect during post-dietary change assessment using ecological momentary assessments (EMA). | Through study completion, an average of 1 month
  Negative Affect is measured by asking participants to self-report affect (e.g., irritability, depression) on their smart phones throughout the day during pre and post dietary change. Participants are asked to give ratings of their current feelings / emotions and to provide contextual information (location, environment, etc.). Response options are a 5 points scale with extreme ends of scale marked as "strongly disagree" and "strongly agree". Changes in ratings from pre dietary change to post dietary change within subjects will be used for analyses
Increase in negative affect during post-dietary change assessment using Profile of Mood Scale (POMS). | Through study completion, an average of 1 month
  Profile of Moods Scale - Abbreviated (POMS) is a well validated, self - report scale of affect. The POMS is used to measure daily global affect. The POMS asks about current feelings / emotions. Response options are "not at all" "a little" "moderate" "quite a bit" and "extremely." Participants are asked to complete these measures daily during pre and post dietary change. Change in self-report responses on the POMS at pre dietary change compared to post dietary change will be used for analyses.
Increase in stress reactivity during post-dietary change using the Positive and Negative Affect Scale (PANAS) as an indicator of negative affect during a stress - exposure task. | Through study completion, an average of 1 month
  Participants will complete a stress task during pre and post dietary change. Food cue reactivity symptoms are measured by asking participants to complete the Positive and Negative Affect Scale (PANAS) which asked about current feeling / emotions. Response options are "very slightly / not at all" "a little" "moderately" "quite a bit" or "extremely." Participants are asked to complete these measures before and after completing a stress exposure task during the pre and post dietary change. The magnitude of change in self - report responses in negative affect in response to the stress task on the PANAS at pre dietary change compared to post dietary change will be used for analyses.
Increased propensity to experience food craving using ecological momentary assessment (EMA). | Through study completion, an average of 1 month
  Food cravings are measured by asking participants to self-report food cravings and to provide contextual information (location, environment, etc.) on their smart phones throughout the day. Response options are a 5 points scale with extreme ends of scale marked as "strongly disagree" and "strongly agree". The magnitude of change in cravings ratings from pre dietary change to post dietary change within subjects will be used for analyses.
Increased propensity to experience food craving using the Food Craving Questionnaire (FCQ - S). | Through study completion, an average of 1 month
  Food cravings are measured by asking participants to complete the Food Craving Questionnaire (FCQ-S) which is a validated measure of current food cravings. Response options are "Strongly Disagree" "Disagree" "Neutral" "Agree" or "Strongly Agree." Participants are asked to complete these measures daily during the pre and post dietary change. Change in self - report responses on the daily report FCQ-S at pre dietary change compared to post dietary change will be used for analyses.
Increased propensity to experience food craving in response to a cue reactivity task using the Food Craving Questionnaire (FCQ - S). | Through study completion, an average of 1 month
  Participants will be shown commercial advertisement videos for highly processed foods during the pre and post dietary change. Food cravings are measured by asking participants to complete the Food Craving Questionnaire (FCQ-S) which is a validated measure of current food cravings. Response options are "Strongly Disagree" "Disagree" "Neutral" "Agree" or "Strongly Agree." The magnitude of change is self - report craving on this measure during pre-dietary change compared to post dietary change will be used for analyses.

SECONDARY OUTCOMES:
Increased hunger in response to cue - reactivity task using subjective hunger measure. | Through study completion, an average of 1 month
  Participants will be shown commercial advertisement videos for highly processed foods during the pre and post dietary change. Participant's subjective craving will be measured on a scale of 0 to 100. Change is self - report responses on this hunger self - report measures during pre-dietary change compared to post dietary change will be used for analyses.
Increased craving in response to cue reactivity task using subjective craving measure. | Through study completion, an average of 1 month
  Participants will be shown commercial advertisement videos for highly processed foods during the pre and post dietary change. Participant's subjective hunger will be measured on a scale of 0 to 100. Change is self - report responses on these self - report measures during pre-dietary change compared to post dietary change will be used for analyses.
Increased hunger in response to stress exposure task using subjective measure of hunger. | Through study completion, an average of 1 month
  Participants will complete a stress task during pre and post dietary change. Participants will listen to a personalized stress script foods during the pre and post dietary change. Participant's subjective hunger will be measured on a scale of 0 to 100. Change is self - report hunger on this self - report measures during pre-dietary change compared to post dietary change will be used for analyses.
Increased craving in response to stress exposure task using subjective measure of craving. | Through study completion, an average of 1 month
  Participants will complete a stress task during pre and post dietary change. Participants will listen to a personalized stress script foods during the pre and post dietary change. Participant's subjective craving will be measured on a scale of 0 to 100. Change is self - report responses on these self - report measures during pre-dietary change compared to post dietary change will be used for analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Gearhardt, Ph.D, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported will be de-identified and shared.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal will be able to access data to achieve aims outlined in the approved proposal. Proposals should be directed to agearhar@umich.edu to gain access. Data requestors will need to sign a data access agreement. Data will be stored by the research team for 5 years.